CLINICAL TRIAL: NCT05976815
Title: Improving Response to Chemotherapy by Adding Physical Exercise in the Neoadjuvant Setting of Breast Cancer Patients - The KEYMOVE Randomized Controlled Trial
Brief Title: Improving Response to Chemotherapy by Adding Physical Exercise in the Neoadjuvant Setting of Breast Cancer Patients
Acronym: KEYMOVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Institute of Maia (Other)
Collaborators: Aveiro University (Other); Centro Hospitalar de Vila Nova de Gaia/Espinho (Other); Associacao de Investigacao de Cuidados de Suporte em Oncologia (Other); University of Maia (Other)
Responsible Party: Principal Investigator, Alberto Alves, Principal Investigator, University Institute of Maia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: keymove
Record Dates: First submitted 2023-06-06; First posted 2023-08-04 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Neoadjuvant Chemotherapy; Physical Exercise; Pathologic Complete Response; Immune System
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Pathologic Complete Response

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group will receive neoadjuvant chemotherapy alone (standard of care).
- Experimental Group (Experimental): The experimental group will receive neoadjuvant chemotherapy (standard of care) in conjunction with an exercise intervention. The exercise intervention will be implemented concurrently for the full duration of the neoadjuvant chemotherapy treatment.
  Interventions: Behavioral: Combined Aerobic and Resistance Exercise

INTERVENTIONS:
Behavioral: Combined Aerobic and Resistance Exercise — Apart from the neoadjuvant chemotherapy treatment (standard of care), participants allocated to the experimental group will additionally participate in a supervised physical exercise program that comprises 3 weekly sessions during the months that the patient is undergoing chemotherapy treatment. Each 75-minute session will comprise a 10-minute warm up, 30 minutes of strength training involving exercise for the major muscle groups, 30 minutes of aerobic training at 40-89% of heart rate reserve and a 5-minute cool down.
  Arms: Experimental Group

SUMMARY:
One of the recommended treatments for breast cancer is neoadjuvant chemotherapy (NCT), however, only 20% of the patients subject to this therapy present pathologic complete response (pCR). If exercise-induced tumour size reductions observed in preclinical studies translates to humans, physical training could emerge as a way of increasing rates of pCR to NCT, which would be a valuable clinical achievement. The present randomized controlled trial primary aim is to assess the impact of a physical exercise intervention the NCT efficacy. Following a parallel-arm design, 86 women with primary BC will be allocated 1:1 to a NCT + exercise (experimental) or NCT alone (control) group. The primary outcome is the rate of pCR in each group. Secondary outcomes include treatment tolerability and compliance, tumour infiltrating lymphocytes, ki67, immune, inflammatory, matricellular and myogenic markers, physical fitness, accelerometry, quality of life and body composition.

ELIGIBILITY:
Inclusion Criteria:

1. being female gender;
2. age equals or greater than 18 years old;
3. having a newly diagnosed histologically confirmed breast carcinoma IA-IIIC;
4. planned to receive neoadjuvant chemotherapy with anthracyclines or taxanes, that might be associated to anti-HER2 drugs;
5. being followed by the oncology department of the CHVNG/E;
6. medical oncologists consents the practice of physical exercise;
7. the patient is capable of providing written informed consent;
8. the participant accepts to be allocated to the control or experimental group, according to the randomization.

Exclusion Criteria:

1. previous cancer diagnostic;
2. evidence of synchronous oncologic disease;
3. physical or psychiatric contraindication to the practice of physical exercise.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response | Post-intervention / Post-treatment. After neoadjuvant chemotherapy, and after surgery. Up to 33 weeks post-baseline.
  Pathological response as the primary outcome will be assessed by a blinded pathologist from the tumour surgical specimens after the breast surgery (post-intervention) and will be defined as complete, partial or no response. Besides pathological complete response (defined as ypT0/ypN0), groups will be compared as those with response (complete or partial) versus those with no response. The residual cancer burden which quantifies residual disease after NAC (post-intervention) will also be assessed.

SECONDARY OUTCOMES:
Treatment Tolerance - clinically assessed. | From baseline (week 0) until the end of chemotherapy, an average of 26 weeks.
  Number of participants with clinically assessed treatment-related adverse events. Will be assessed according to the Common Terminology Criteria for Adverse Events v5.0. The scale uses a minimal value of 1 and a maximal value of 5 to grade each adverse event, with higher scores representing worse outcomes.
Treatment Tolerance - patient reported. | From baseline (week 0) until the end of chemotherapy, an average of 26 weeks.
  Number of participants with patient-reported adverse events. Will be assessed using the Patient reported outcomes version of the Common Terminology Criteria for Adverse Events v1.0 questionnaire. The scale uses a minimal rating 0 and a maximal rating of 4 to grade each adverse event, with higher scores representing worse outcomes.
Chemotherapy Relative Dose Intensity | From baseline (week 0) until the end of chemotherapy, an average of 26 weeks.
  Chemotherapy relative dose intensity will be calculated by the following formula: (Delivered dose intensity / Standard dose intensity) x 100%, where Delivered dose intensity = (Delivered total dose, in mg/m2)/(actual time to complete chemotherapy with imputation for missed cycles, in days) and Standard Dose Intensity = (Standard total dose, in mg/m2)/(standard time to complete chemotherapy, in days).
Number of Chemotherapy Dose Reductions | From baseline (week 0) until the end of chemotherapy, an average of 26 weeks.
  Number of patients that had to reduce the dose of chemotherapy from the dose of chemotherapy initially prescribed (standard dose intensity).
Number of Chemotherapy Delays | From baseline (week 0) until the end of chemotherapy, an average of 26 weeks.
  Number of patients that had to delay a cycle of chemotherapy, in comparison to what had initially been prescribed (standard dose intensity).
Number of Chemotherapy Early Discontinuations | From baseline (week 0) until the end of chemotherapy, an average of 26 weeks.
  Number of patients that had to interrupt chemotherapy before the standard dose had been administrated.
Percentage of Tumor Infiltrating Lymphocytes | At baseline (week 0) and post-intervention (after an average of 30 weeks from study enrolment).
  Assessed at Histology Slides. Intratumoral and stromal infiltrating lymphocyte (TIL) population will be assessed in tumour biopsies (at baseline) and surgical resection specimens collected from the post-neoadjuvant chemotherapy surgery (post-intervention). This will be used to compute intratumoral and stromal TIL's score, recorded as the percentage of TIL's on the analysed area. Only stromal TIL ́s will be quantified in patients with complete pathological response.
Percentage of Tumor Ki67 | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  Assessed at Histology Slides. Ki67 will be assessed in tumour biopsies (at baseline) and surgical resection specimens collected from the post-neoadjuvant chemotherapy surgery (post-intervention).
Percentage of Cytotoxic T Cells on Peripheral Blood | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  Flow cytometry will be the method used to assess the number of CD3+CD8+ (cytotoxic T cells) on peripheral blood lymphocytes.
Percentage of Natural Killer T Cells on Peripheral Blood | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  Flow cytometry will be the method used to assess the number of CD3+CD56+ (natural killer T cells) on peripheral blood lymphocytes.
Percentage of T Helper Cells on Peripheral Blood | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  Flow cytometry will be the method used to assess the number of CD3+CD4+ (T helper cells) on peripheral blood lymphocytes.
Plasma IFN-gamma levels | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  The enzyme-linked immunosorbent assay method will be used to identify the concentration of the cytokine IFN-gamma on plasma.
Plasma TNF-alpha levels | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  The enzyme-linked immunosorbent assay method will be used to identify the concentration of the cytokine TNF-alpha on plasma.
Plasma Irisin Levels | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  The enzyme-linked immunosorbent assay method will be used to identify the concentration of the hormone Irisin on plasma.
Plasma SPARC levels | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  The enzyme-linked immunosorbent assay method will be used to identify the concentration of the protein SPARC on plasma.
Plasma Decorin Levels | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  The enzyme-linked immunosorbent assay method will be used to identify the concentration of the protein Decorin on plasma.
Plasma Oncostatin M Levels | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  The enzyme-linked immunosorbent assay method will be used to identify the concentration of the cytokine Oncostatin-M on plasma.
Distance traveled in the 10 meter-incremental shuttle walk test | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  As an indicator of cardiorespiratory fitness, the number of meters that the participant is able to walk/run in the 10 meter-incremental shuttle walk test will be assessed.
Maximal METS reached during a cardiopulmonary exercise test | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  The participant will be subjected to a maximal incremental conventional cardiopulmonary exercise test on a treadmill. The maximal intensity the participant is able to attain in this assessment will be recorded in METS.
Number of repetitions performed in the 30 second sit-to-stand test | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  The 30 second sit-to-stand test will be used to assess lower limb dynamic muscular strength. The maximal number of repetitions the participant is able to perform in the 30 second sit-to-stand test will be recorded.
Maximal Isometric Handgrip Strength | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  The maximal force (in kilograms) the participant is able to produce in an isometric handgrip test will be recorded, using a hand dynamometer.
Maximal Isometric Quadriceps Strength | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  The maximal force (in kilograms) the participant is able to produce in an isometric strength test for the quadriceps muscle will be recorded using a load cell. Additionally, the time to maximal strength (in seconds) will also be recorded.
Weekly time time spent in light, moderate and vigorous physical activities and sedentary behaviours. | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  Assessed by accelerometry over a period of seven days, the time (in minutes) that the participants spend in light, moderate and vigorous physical activity will be recorded. Additionally, the time (in minutes) spent in sedentary behaviours will also be recorded.
Health-Related Quality of Life | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  The questionnaires European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (version 1.0) and the Breast 23 Questionnaire (version 1.0) will be implemented to assess cancer-related quality of life. The final scores will range from 0 to 100, with higher scores on the functional scales representing a high level of functioning and higher scores on the symptom scales implying a stronger symptom burden.
Total Body Weight | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  Using bioimpedance, the participants' total body weight, in kilograms, will be assessed with the lightest clothes possible.
Total Body Skeletal Muscle Mass | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  Using bioimpedance, the participants' total body skeletal muscle mass, in kilograms, will be assessed.
Total Body Fat | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  Using bioimpedance, the participants' total body fat, in kilograms, will be assessed.
Body Mass Index | At baseline (week 0) and post-intervention (after an average of 30 weeks post study enrolment).
  Using weight and height, these parameters will be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Nuno Rato, MSc, Principal Investigator — University of Maia
Locations (1):
- Centro Hospitalar Vila Nova Gaia e Espinho, Vila Nova de Gaia, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No